CLINICAL TRIAL: NCT03832959
Title: Evaluation of Esophageal Damage During Conventional Pulmonary Vein Ablation Procedures and Potential Strategies to Protect the Esophagus. Pilot Study.
Brief Title: Esophageal Damage Protection During Pulmonary Vein Ablation. Pilot Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-ABL-2018-55
Record Dates: First submitted 2019-01-16; First posted 2019-02-06 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation; Catheter Ablation; Esophageal Fistula; Esophageal Diseases; Arrhythmias, Cardiac
MeSH Terms: conditions — Atrial Fibrillation; Esophageal Fistula; Esophageal Diseases; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Patients referred for catheter ablation of atrial fibrillation (either cryoablation or radiofrequency ablation (1/1)) will be randomized to either receive or not (1/1) an esophageal temperature adjustment EnsoETM device, to evaluate its role for esophageal protection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Non esophageal protection (No Intervention): Patients in this group will undergo a first atrial fibrillation catheter ablation procedure with pulmonary vein isolation to study esophageal lesions. The esophageal protection probe will not be used.
- Esophageal protection (Experimental): Patients in this group will undergo a first atrial fibrillation catheter ablation procedure with pulmonary vein isolation, using the esophageal protection probe EnsoETM
  Interventions: Device: EnsoETM

INTERVENTIONS:
Device: EnsoETM — The EnsoETM is a device with a esophageal probe that can provide temperature adjustment
  Arms: Esophageal protection

SUMMARY:
Catheter ablation of atrial fibrillation with electrical isolation of the pulmonary veins in the left atrium carries risk of esophagus thermal lesion. EnsoETM is a device . This study evaluates the benefit of using the EnsoETM, a device device for esophageal temperature adjustments, during catheter ablation of atrial fibrillation. Half of participants will undergo esophageal temperature adjustment during pulmonary vein catheter ablation, while the other half will undergo catheter ablation with no esophageal temperature adjustment.

DETAILED DESCRIPTION:
1. THEORETICAL FRAMEWORK. APPROACH TO THE PROBLEM

Background and justification

Atrial fibrillation is the most common type of heart arrhythmia. Electrical isolation of the pulmonary veins in the left atrium with ablation is standard therapy in the invasive treatment of atrial fibrillation. One of the risks of this intervention is thermal lesion of the esophagus, since it is in contact with the posterior wall of the left atrium. The energy applied for electrical isolation via either radiofrequency or cryotherapy can cause thermal lesions due to proximity with the esophagus and the vagus nerve/parasympathetic nervous system of the upper digestive tract. The incidence is not well established and data in the existing scarce publications show a very wide range, from 3 to 60%, according to the definition and means of the study used. The most recent systematic studies show values around 40-50%. The lesions observed vary in degree, from erythema or minor erosion to ulcers of the esophageal mucosa, including local hematomas, spasms, and esophageal/gastric motility disorders and even atrial-esophageal fistula, the extreme consequence of thermal esophageal lesion; the incidence of the latter is low (0.25%), but it has an elevated mortality. The best examination to diagnose and evaluate these lesions in all phases is upper digestive endoscopy or fibro esophagogastroscopy. Although it is routine in digestive services throughout the world, enabling the direct visualization and characterization of lesions, this technique is not performed systematically after ablation procedures, which explains the contradictory data in the literature.

Likewise, the possible long-term consequences of minor lesions are unknown, which, in a large number of patients are totally asymptomatic. For this reason, it cannot be ignored that acute tissue damage, however minimal, could lead to future changes in the form of late onset chronic esophageal pathology. The incidence and magnitude of esophageal involvement has been directly related to the ablation technique and protocol. Most available studies have been carried out in centers with ablation protocols that are significantly more aggressive than those used in our care facility. For this reason, the investigators do not have reliable data regarding the size of the problem in our center, which could present some differential characteristics.

To date, the prevention of these esophageal lesions has entailed: limits in the energy applied on the posterior wall of the left atrium (less power or shorter application time); monitoring of the luminal esophageal temperature during radio frequency or cryotherapy applications; stopping application early if certain temperatures considered risky were reached. However, the success of luminal esophageal temperature monitoring in preventing lesions varies widely, given that the temperature probes are very thin with respect to the total diameter of the esophagus, their position varies with respect to the cardiac tissue treated, and contact with the esophageal mucosa is inconstant. In fact, it has been reported that the temperature probes used for monitoring can contribute to increasing thermal lesions, given that their metal elements can boost direct heating/cooling of the tissue and make the lesion larger and last longer. In fact, the incidence of esophageal lesions is very similar, independent of the use of the temperature probe, or if it is a single or multi-sensor. Another controversial aspect of these temperature probes is that their use can lead to - at least potentially and in pursuit of safety - shorter, limited applications, which could cause incomplete non-transmural lesions and hamper the correct treatment of patients, thereby becoming a factor that increases the recurrence of atrial fibrillation. In addition, these probes should be deployed during the procedure so they are as close as possible to the application site (right or left veins depending on the time), which increases the procedure and fluoroscopy time, with consequent risks for both the patient and the medical team. All these limitations, together with significant economic cost overruns have meant that the use of this approach in our care facilities has been minimal and only for research purposes.

Even if the possible long-term consequences of esophageal lesions are minimal, studying new strategies for esophageal protection that are easy to implement and do not affect the efficacy of ablation procedures is of great clinical and scientific interest. In this context, there is a plan to use the probes to regulate and maintain patient temperature in prolonged surgeries or critical units as a method of esophageal protection during ablation. Multiple clinical studies have demonstrated the efficacy and safety of these probes in different medical/surgical areas. In particular, they are indicated to minimize the neurological damage associated with heart attacks through the induction of therapeutic hypothermia. They are also indicated to reduce the temperature of patients with malignant hyperthermia, to prevent unexpected peri-operative hypothermia, and to reduce elevated intracranial pressure.

The prevention of esophageal lesions via temperature control (local cooling of the esophagus when radiofrequency is used or heating when cryotherapy is used, thanks to various probe configurations) has been investigated with mathematical models, preclinical models, and in the clinical field in a preliminary way. Data are available that demonstrate its efficacy in this approach, although with limitations in the number of cases and the systems used. In most of these studies, prototypes of anterior probes were used, which are difficult to place and require changes in the work routine, which has made the expansion of devices using this approach more difficult up to now.

The appearance of a new, easier-to-use device for esophageal temperature adjustments (EnsoETM, Attune Medical, Chicago, Illinois, USA) when managing patient temperature for a large variety of needs has facilitated the reintroduction of this therapeutic option.

The EnsoETM, made by Attune Medical, received its CE mark in Europe in 2014, with an expanded indicated use of up to 120 hours in 2016 and a CE mark for its use with the Altrix system by Stryker® in 2017. (CE certificate attached.) The EnsoETM is used as part of treatment to obtain therapeutic hypothermia during the management of a heart attack. It is also used in the treatment of hyperthermia, the prevention of unexpected peri-operative hypothermia, and the reduction of elevated intracranial pressure.

The device is situated in the esophagus like a standard orogastric sensor. A multi-channel cylindrical silicone tube connected to a closed water circuit allows the surrounding tissue to be warmed or cooled according to the need or desired temperature. This effect is achieved through the transfer of heat via conduction through the esophagus and by convection through the device. One must keep in mind that the posterior wall of the left atrium is in close contact with the esophagus and the modular effect of the temperature therefore also acts on the wall of the atrium.

The EnsoETM is designed to use the high-blood-flow surroundings of the esophagus and achieve high heat-exchange performance. In addition, the EnsoETM has a distal end that reaches the stomach and allows it to be decompressed, avoiding distension of the esophagus, which ensures good contact between the device and the esophageal mucosa, thereby maximizing the transfer of heat between the device and the patient. The EnsoETM is composed of standard medical-grade silicone, and is generally similar in shape and size to gastric probes and other devices that are routinely situated in the esophagus (esophagogastroduodenoscopes, transesophageal echocardiogram probes, Ewald tubes, etc.). It is also smaller than other more aggressive devices (the EnsoETM measures approximately 1/3 the size of the Sengstaken-Blakemore tube used to treat esophageal varices).

The preliminary data available show that the use of probes that regulate the esophageal temperature would allow the mucosa of thermal lesions to be protected, thereby reducing and preventing lesions on this level during the fibrillation ablation treatment. However, it is not known whether the modulation of esophageal temperature or contact with the atrial wall affect the efficacy of the actual lesions induced on the atrium and therefore on the success of the ablation procedure.

Hypothesis

General hypothesis:

Esophageal protection probes allow the deleterious effects of pulmonary vein ablation to be counteracted on the wall of the esophagus.

Secondary hypotheses:

1. The incidence of esophageal lesions in our setting, in which a conservative approach is applied to the ablation of pulmonary veins, is low but not insignificant.

2 The use of esophageal protection probes allows the incidence of esophageal lesions to be decreased.

3 The use of esophageal protection probes does not alter the clinical result of the pulmonary vein ablation procedure.

2. GENERAL AND SPECIFIC OBJECTIVES:

Main objective:

Assess the role of esophageal protection probes during pulmonary vein ablation procedures.

Secondary objectives

1. Assess the incidence of esophageal lesions in our setting.
2. Assess if the use of a probe for esophageal protection reduces the incidence of esophageal lesions.
3. Assess if the use of esophageal protection probes alters the clinical result of the pulmonary vein ablation procedure.

3. METHODS:

Study design

The investigators propose a prospective pilot study to assess the incidence of esophageal lesions following a pulmonary vein ablation procedure in our care center in which a conservative approach is used to apply the energy. In addition, in a limited number of patients, the study aims to assess the effect of an esophageal protection probe on the occurrence of thermal lesions and the results of the ablation.

The study protocol will be carried out under the directives of the Institutional Ethics Committee in the Hospital de la Santa Creu i Sant Pau.

Patients referred for catheter ablation of atrial fibrillation (either cryoablation or radiofrequency ablation (1/1)) will be randomized to either receive or not (1/1) an esophageal temperature adjustment EnsoETM device, to evaluate its role for esophageal protection.

Ablation procedure:

All patients included in the study will be subject to an ablation procedure following the standard guidelines in our center with no modification, where the investigators carry out the procedures under general anesthesia. Instead of using a conventional orogastric probe, the patients in the probe-evaluation group will systematically use the probe protecting against thermal lesions with no other variation.

Use of the EnsoETM esophageal probe:

Placement of the EnsoETM will follow standard recommendations according to the instructions, which are similar to recommendations for inserting a transesophageal echocardiogram probe (routine procedure in some centers to guide the transseptal puncture) or the orogastric aspiration probe during surgical procedures. The EnsoETM will be connected to the appropriate console (Meditherm, Blanketrol, or Altrix). The configuration will be adjusted according to the ablation technique (cryoablation or radiofrequency ablation). If radio frequency is used, before beginning the ablation of the left posterior wall, the heat exchanger connected to the EnsoETM will be adjusted to a cooling mode (5°C), with ablation beginning at least 1 min after the circulating water reaches a temperature of 5°C. If cryoablation is used, before beginning the application, the heat exchanger connected to the EnsoETM will be adjusted to a heating mode (45°C), with cryoablation beginning at least 1 min after the circulating water reaches a temperature of 45°C.

Esophagogastroscopy:

An esophagogastroscopy will be done on all patients, a day later after the catheter ablation, following the usual guidelines of the Gastroenterology Service. Local anesthesia will be used with superficial sedation following a 12-hour fast. Basal anticoagulant treatment will be maintained without any precise antibiotic prophylaxis. The gastroenterologist will provide a report on the procedure, classifying the findings in agreement with Zargar's criteria, assessing them qualitatively as light, moderate, or serious. Special focus will be placed on the anterior zone of the esophagus at the level of the left atrium, which is where the energy (radio frequency or cryoablation) is applied during the procedure.

Monitoring:

The usual treatment and controls will both be followed unless the gastroenterologist changes the recommendations due to the endoscopy findings. Follow-up visits will be made at 1, 3, 6, and 12 after the procedure to assess the presence of cardiological and gastrointestinal symptoms.

Study population. The population will consist of patients subjected to their first pulmonary vein ablation procedure in the left atrium to treat atrial fibrillation.

Definition of variables

1. Demographic variables: age, gender, weight, and height
2. Clinical variables: cardiovascular risk factors, atrial fibrillation factors (alcohol, sleep apnea, obesity, …), previous atrial fibrillation arrhythmia, history of gastrointestinal pathology (reflux, esophagitis, gastritis, H Pylori infection, …), history of cardiological pathology (basic structural cardiomyopathy: ischemic, valvular, hypertensive, diameter and volume of the left atrium, ejection fraction, …).
3. Family history of early atrial fibrillation (<40 years).
4. Previous pharmacological treatment: especially anti-arrhythmia, anticoagulant and anti-secretion or gastric protector (indication, dosage, time, and administration route).
5. Effectiveness of pulmonary vein isolation.
6. Radio-physical variables of the ablation (number of applications, duration of application, maximum or minimum temperature, power (W), ablation index per region (anterior, posterior).
7. Duration of procedure: fluoroscopy, catheterization in the left atrium.
8. Clinical or electrical efficacy. Recurrence of arrhythmia (palpitations, ECG, or Holter monitor)
9. Esophageal lesions per Zargar endoscopy classification
10. Adverse clinical events

    * Dysphagia: the patient relates difficulty swallowing for more than 24 hours after the use of the device; diagnosed via modified barium swallow study, videofluoroscopic swallow study, or related directly by the patient.
    * Odynophagia: the patient relates pain when swallowing for more than 24 hours after the use of the device; diagnosed via the patient's subjective feelings.
    * Esophageal lesion not due to ablation: evidence of traumatic lesions or other esophageal lesions diagnosed by a gastroenterologist.

Sample size and strength Given that the incidence of esophageal lesions in recent studies was estimated to be 40-50%, and a reduction of 20% was calculated in the appearance of lesions with the use of the probe compared to control conditions (without modification of the esophageal temperature), with a power of 80% and an alpha error of 0.05. A necessary sample size of 28 patients was specified for each of the techniques used (radio frequency and cryoablation).

Method. Sources of information The information gathered throughout the study will be collected in an encrypted database designed and built specifically for the study. Atrial fibrillation ablation is a common technique in our center, with more than 100 procedures performed annually.

Data management and analysis Statistical analysis will be carried out with the statistics program SPSS, version 25.0 (IBM Corporation). The continuous variables will be expressed as an average and standard variation or medians and interquartile range, depending on whether the distribution is statistically different from a normal distribution. Qualitative variables will be presented as numbers and percentages. To study the relationship between qualitative variables, the chi-squared test (X2) will be used; Fisher's exact test will be used for variables that do not follow a normal distribution. The quantitative variables will be compared using Student's t-test if two groups are compared; analysis of variance (ANOVA) will be used for more than two groups. If the quantitative variables do not follow a normal distribution, non-parametric tests will be used: the Mann-Whitney U-test for two groups or the Kruskal-Wallis test for more than two groups. The correlation between the variables will be studied using the Pearson or Spearman tests, depending on whether the distribution is normal or not. Differences with a p-value of 0.05 or higher will be considered significant.

The only significant change with respect to usual practice is that an upper digestive endoscopy will be performed on all patients included. However, this activity is not expected to lead to a change in the length of admission or in the treatment administered. Although it is a new element, the introduction of the probe is not expected to lead to significant changes, since all patients are intubated in the usual way and, based on need, a nasogastric probe of reduced size will simultaneously be introduced in the same way as the study probe to avoid gastric distension.

5. WORK PLAN (tasks, benchmarks and timeline of the study): Month 1 Development of the protocol. Editing of study materials. Design of the database. Researcher meeting to resolve doubts. Preparation of logistical aspects to begin the study.

Month 2 Presentation to the Research Ethics Committee. Months 3-12 Beginning of the study. Dissemination of the services involved (cardiology, anesthesiology, gastroenterology). Data collection and entry.

Months 12-18 Data cleaning and analysis. Researcher meeting to resolve doubts and close the study. Drafting of the final report. Drafting of a manuscript to publish the results.

Duration: 18 months

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (older than 18 years of age) subjected to their first pulmonary vein isolation procedure with a catheter or balloon.

Exclusion Criteria:

* Patients with known esophageal deformity or evidence of esophageal trauma (for example, history of esophagectomy, previous swallowing disorders, achalasia, etc.)
* Patients with known ingestion of acidic or caustic poison in the previous 24 hours.
* Patients weighing less than 40 kg.
* Patients who know they are pregnant.
* Patients under chronic daily treatment with an proton pump inhibitor or any gastrointestinal acid suppressant.
* Patients under 18 years of age.
* Patients who have not signed the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Presence of esophageal damage | 1 day
  Presence of esophageal lesions will be determined after ablation using esophagogastroscopy.
Severity of esophageal damage | 1 day
  Degree of esophageal lesions will be determined after ablation using esophagogastroscopy. Degree of esophageal lesions severity will be determined according to the Zargar endoscopy classification (0, I, IIa, IIb, IIIa, IIIb, IV)
Presence of esophageal damage | <48 hours
  Presence of esophageal lesions will be determined after ablation using magnetic resonance imaging

SECONDARY OUTCOMES:
Recurrence of atrial fibrillation | 1 year
  Recurrence of atrial fibrillation after catheter ablation will be determined in the follow-up:
  1. clinically, as episodes with high clinical suspicion of being atrial fibrillation despite no ECG documentation
  2. documented in ECG or in 24-hours holter monitoring, and defined as an episode lasting more than 30 seconds. 24-hours holter monitoring will be performed 3, 6 and 12 months after catheter ablation

CONTACTS AND LOCATIONS:
Overall Officials: Jose Maria Guerra Ramos, MD PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
There is no IPD sharing plan

REFERENCES:
- [Background] Tzou WS, Russo AM. Luminal esophageal temperature monitoring for the prevention of esophageal injury during left atrial ablation: LET it be? J Cardiovasc Electrophysiol. 2013 Sep;24(9):965-7. doi: 10.1111/jce.12198. Epub 2013 Jul 19. No abstract available. PMID 23869691
- [Background] Nair GM, Nery PB, Redpath CJ, Lam BK, Birnie DH. Atrioesophageal fistula in the era of atrial fibrillation ablation: a review. Can J Cardiol. 2014 Apr;30(4):388-95. doi: 10.1016/j.cjca.2013.12.012. Epub 2013 Dec 20. PMID 24582720
- [Background] Liu E, Shehata M, Liu T, Amorn A, Cingolani E, Kannarkat V, Chugh SS, Wang X. Prevention of esophageal thermal injury during radiofrequency ablation for atrial fibrillation. J Interv Card Electrophysiol. 2012 Oct;35(1):35-44. doi: 10.1007/s10840-011-9655-0. Epub 2012 Jun 21. PMID 22717996
- [Background] 10.5935/abc.20160078
- [Background] Tschabrunn CM, Silverstein J, Berzin T, Ellis E, Buxton AE, Josephson ME, Anter E. Comparison between single- and multi-sensor oesophageal temperature probes during atrial fibrillation ablation: thermodynamic characteristics. Europace. 2015 Jun;17(6):891-7. doi: 10.1093/europace/euu356. Epub 2015 Mar 15. PMID 25777771
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation: Executive summary. J Arrhythm. 2017 Oct;33(5):369-409. doi: 10.1016/j.joa.2017.08.001. Epub 2017 Sep 15. No abstract available. PMID 29021841
- [Background] Halm U, Gaspar T, Zachaus M, Sack S, Arya A, Piorkowski C, Knigge I, Hindricks G, Husser D. Thermal esophageal lesions after radiofrequency catheter ablation of left atrial arrhythmias. Am J Gastroenterol. 2010 Mar;105(3):551-6. doi: 10.1038/ajg.2009.625. Epub 2009 Nov 3. PMID 19888201
- [Background] Knopp H, Halm U, Lamberts R, Knigge I, Zachaus M, Sommer P, Richter S, Bollmann A, Hindricks G, Husser D. Incidental and ablation-induced findings during upper gastrointestinal endoscopy in patients after ablation of atrial fibrillation: a retrospective study of 425 patients. Heart Rhythm. 2014 Apr;11(4):574-8. doi: 10.1016/j.hrthm.2014.01.010. Epub 2014 Jan 10. PMID 24418167
- [Background] Vaezi MF, Pandolfino JE, Vela MF. ACG clinical guideline: diagnosis and management of achalasia. Am J Gastroenterol. 2013 Aug;108(8):1238-49; quiz 1250. doi: 10.1038/ajg.2013.196. Epub 2013 Jul 23. PMID 23877351
- [Background] Leite LR, Santos SN, Maia H, Henz BD, Giuseppin F, Oliverira A, Zanatta AR, Peres AK, Novakoski C, Barreto JR, Vassalo F, d'Avila A, Singh SM. Luminal esophageal temperature monitoring with a deflectable esophageal temperature probe and intracardiac echocardiography may reduce esophageal injury during atrial fibrillation ablation procedures: results of a pilot study. Circ Arrhythm Electrophysiol. 2011 Apr;4(2):149-56. doi: 10.1161/CIRCEP.110.960328. Epub 2011 Feb 15. PMID 21325208
- [Background] Carroll BJ, Contreras-Valdes FM, Heist EK, Barrett CD, Danik SB, Ruskin JN, Mansour M. Multi-sensor esophageal temperature probe used during radiofrequency ablation for atrial fibrillation is associated with increased intraluminal temperature detection and increased risk of esophageal injury compared to single-sensor probe. J Cardiovasc Electrophysiol. 2013 Sep;24(9):958-64. doi: 10.1111/jce.12180. Epub 2013 Jun 7. PMID 23746064
- [Background] Hornero F, Berjano EJ. Atrial ablation and esophageal injury: comments on an experimental study. J Thorac Cardiovasc Surg. 2006 Jul;132(1):212-3; author reply 213-4. doi: 10.1016/j.jtcvs.2006.02.040. No abstract available. PMID 16798355
- [Background] Deneke T, Bunz K, Bastian A, Pasler M, Anders H, Lehmann R, Meuser W, de Groot JR, Horlitz M, Haberkorn R, Mugge A, Shin DI. Utility of esophageal temperature monitoring during pulmonary vein isolation for atrial fibrillation using duty-cycled phased radiofrequency ablation. J Cardiovasc Electrophysiol. 2011 Mar;22(3):255-61. doi: 10.1111/j.1540-8167.2010.01916.x. Epub 2010 Oct 11. PMID 20958829
- [Background] Hegazy AF, Lapierre DM, Butler R, Martin J, Althenayan E. The esophageal cooling device: A new temperature control tool in the intensivist's arsenal. Heart Lung. 2017 May-Jun;46(3):143-148. doi: 10.1016/j.hrtlng.2017.03.001. Epub 2017 Apr 11. PMID 28410771
- [Background] Wayne, M. The Esophageal Cooling Device: A New Way to Achieve Targeted Temperature Management. J Cardiol & Cardiovasc Ther. 5 (1), doi:10.19080/JOCCT.2017.05.555651, (2017).
- [Background] Markota A, Kosir AS, Balazic P, Zivko I, Sinkovic A. A Novel Esophageal Heat Transfer Device for Temperature Management in an Adult Patient with Severe Meningitis. J Emerg Med. 2017 Jan;52(1):e27-e28. doi: 10.1016/j.jemermed.2016.07.086. Epub 2016 Sep 19. No abstract available. PMID 27658559
- [Background] Zivko, I., Balazic, P., Markota, A. & Sinkovic, A. in 12th Emirates Critical Care Conference (Dubai, UAE, 2016).
- [Background] Markota A, Fluher J, Kit B, Balazic P, Sinkovic A. The introduction of an esophageal heat transfer device into a therapeutic hypothermia protocol: A prospective evaluation. Am J Emerg Med. 2016 Apr;34(4):741-5. doi: 10.1016/j.ajem.2016.01.028. Epub 2016 Jan 28. PMID 26906333
- [Background] Khan, I. et al. in 14th Annual Neurocritical Care Society Meeting (National Harbor, MD, 2016).
- [Background] Markota A, Kit B, Fluher J, Sinkovic A. Use of an oesophageal heat transfer device in therapeutic hypothermia. Resuscitation. 2015 Apr;89:e1-2. doi: 10.1016/j.resuscitation.2015.01.032. Epub 2015 Feb 7. No abstract available. PMID 25660954
- [Background] Markota, A., Fluher, J., Balazic, P., Kit, B. & Sinkovic, A. Therapeutic hypothermia with esophageal heat transfer device. Resuscitation. 96 138, doi:10.1016/j.resuscitation.2015.09.328, (2015).
- [Background] Hegazy AF, Lapierre DM, Butler R, Althenayan E. Temperature control in critically ill patients with a novel esophageal cooling device: a case series. BMC Anesthesiol. 2015 Oct 19;15:152. doi: 10.1186/s12871-015-0133-6. PMID 26481105
- [Background] Goury A, Voicu S, Deye N. Reply letter to: Targeted temperature management using the "Esophageal Cooling Device" after cardiac arrest (the COOL study): A feasibility and safety study. Resuscitation. 2018 Feb;123:e7-e8. doi: 10.1016/j.resuscitation.2017.12.001. No abstract available. PMID 29306528
- [Background] Primozic KK, Svensek F, Markota A, Sinkovic A. Rewarming After Severe Accidental Hypothermia Using the Esophageal Heat Transfer Device: A Case Report. Ther Hypothermia Temp Manag. 2018 Mar;8(1):62-64. doi: 10.1089/ther.2017.0017. Epub 2017 Sep 21. PMID 28934599
- [Background] Naiman, M. et al. An evaluation of esophageal temperature management in cases longer than 72 hours. Resuscitation. 118 e82, doi:10.1016/j.resuscitation.2017.08.198, (2017).
- [Background] Khan I, Haymore J, Barnaba B, Armahizer M, Melinosky C, Bautista MA, Blaber B, Chang WT, Parikh G, Motta M, Badjatia N. Esophageal Cooling Device Versus Other Temperature Modulation Devices for Therapeutic Normothermia in Subarachnoid and Intracranial Hemorrhage. Ther Hypothermia Temp Manag. 2018 Mar;8(1):53-58. doi: 10.1089/ther.2017.0033. Epub 2017 Dec 13. PMID 29236581
- [Background] Williams D, Leslie G, Kyriazis D, O'Donovan B, Bowes J, Dingley J. Use of an Esophageal Heat Exchanger to Maintain Core Temperature during Burn Excisions and to Attenuate Pyrexia on the Burns Intensive Care Unit. Case Rep Anesthesiol. 2016;2016:7306341. doi: 10.1155/2016/7306341. Epub 2016 Feb 25. PMID 27018074
- [Background] Kalasbail P, Makarova N, Garrett F, Sessler DI. Heating and Cooling Rates With an Esophageal Heat Exchange System. Anesth Analg. 2018 Apr;126(4):1190-1195. doi: 10.1213/ANE.0000000000002691. PMID 29283916
- [Background] Berjano EJ, Hornero F. A cooled intraesophageal balloon to prevent thermal injury during endocardial surgical radiofrequency ablation of the left atrium: a finite element study. Phys Med Biol. 2005 Oct 21;50(20):N269-79. doi: 10.1088/0031-9155/50/20/N03. Epub 2005 Sep 27. PMID 16204868
- [Background] Lequerica JL, Berjano EJ, Herrero M, Hornero F. Reliability assessment of a cooled intraesophageal balloon to prevent thermal injury during RF cardiac ablation: an agar phantom study. J Cardiovasc Electrophysiol. 2008 Nov;19(11):1188-93. doi: 10.1111/j.1540-8167.2008.01229.x. Epub 2008 Jun 4. PMID 18554206
- [Background] Lequerica JL, Berjano EJ, Herrero M, Melecio L, Hornero F. A cooled water-irrigated intraesophageal balloon to prevent thermal injury during cardiac ablation: experimental study based on an agar phantom. Phys Med Biol. 2008 Feb 21;53(4):N25-34. doi: 10.1088/0031-9155/53/4/N01. Epub 2008 Jan 16. PMID 18263938
- [Background] Arruda MS, Armaganijan L, Di Biase L, Rashidi R, Natale A. Feasibility and safety of using an esophageal protective system to eliminate esophageal thermal injury: implications on atrial-esophageal fistula following AF ablation. J Cardiovasc Electrophysiol. 2009 Nov;20(11):1272-8. doi: 10.1111/j.1540-8167.2009.01536.x. Epub 2009 Jun 30. PMID 19572955
- [Background] Tsuchiya T, Ashikaga K, Nakagawa S, Hayashida K, Kugimiya H. Atrial fibrillation ablation with esophageal cooling with a cooled water-irrigated intraesophageal balloon: a pilot study. J Cardiovasc Electrophysiol. 2007 Feb;18(2):145-50. doi: 10.1111/j.1540-8167.2006.00693.x. Epub 2006 Dec 1. PMID 17239114
- [Background] Scanavacca, M. I. et al. in ESC Congress 2007, 1 - 5 September Vol. 28 156 (Vienna, Austria, 2007).
- [Background] Kuwahara T, Takahashi A, Okubo K, Takagi K, Yamao K, Nakashima E, Kawaguchi N, Takigawa M, Watari Y, Sugiyama T, Handa K, Kimura S, Hikita H, Sato A, Aonuma K. Oesophageal cooling with ice water does not reduce the incidence of oesophageal lesions complicating catheter ablation of atrial fibrillation: randomized controlled study. Europace. 2014 Jun;16(6):834-9. doi: 10.1093/europace/eut368. Epub 2014 Jan 26. PMID 24469436
- [Background] Sohara H, Satake S, Takeda H, Yamaguchi Y, Nagasu N. Prevalence of esophageal ulceration after atrial fibrillation ablation with the hot balloon ablation catheter: what is the value of esophageal cooling? J Cardiovasc Electrophysiol. 2014 Jul;25(7):686-92. doi: 10.1111/jce.12394. Epub 2014 Mar 24. PMID 24576252
- [Background] Naiman M, Shanley P, Garrett F, Kulstad E. Evaluation of advanced cooling therapy's esophageal cooling device for core temperature control. Expert Rev Med Devices. 2016 May;13(5):423-33. doi: 10.1080/17434440.2016.1174573. Epub 2016 Apr 15. PMID 27043177
- [Background] Naiman MI, Gray M, Haymore J, Hegazy AF, Markota A, Badjatia N, Kulstad EB. Esophageal Heat Transfer for Patient Temperature Control and Targeted Temperature Management. J Vis Exp. 2017 Nov 21;(129):56579. doi: 10.3791/56579. PMID 29286452
- [Background] Zargar SA, Kochhar R, Mehta S, Mehta SK. The role of fiberoptic endoscopy in the management of corrosive ingestion and modified endoscopic classification of burns. Gastrointest Endosc. 1991 Mar-Apr;37(2):165-9. doi: 10.1016/s0016-5107(91)70678-0. PMID 2032601